CLINICAL TRIAL: NCT02946619
Title: Reducing Psychological Burdens Among Chinese Breast Cancer Survivors
Brief Title: Health Benefits of Expressive Writing Among Chinese Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: American Cancer Society, Inc. (Other); Herald Cancer Association (Other)
Responsible Party: Principal Investigator, Qian Lu, Associate Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MRSGT-10-011-01-CPPB
Record Dates: First submitted 2016-10-21; First posted 2016-10-27 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: Chinese breast cancer survivors; expressive writing
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Condition (No Intervention): Participants in the control group were asked to write for three weeks about facts regarding their cancer and its treatment for three sessions.
- Self-regulation condition (Experimental): For the self-regulation condition, each weekly writing assignment covers a different task. During session one, participants will be asked to write about their deepest feelings and thoughts regarding their experience with breast cancer as well as its impact on their lives; in session two, participants will be asked to write about their coping strategies to deal with stressors associated with the cancer diagnosis and treatment, as well as future plans for coping with cancer-related stressors; and in session three, participants will be asked to write about positive thoughts and feelings regarding their experience with breast cancer.
  Interventions: Behavioral: Self-Regulation Condition
- Enhanced self-regulation condition (Experimental): For the enhanced self-regulation condition, each weekly writing assignment covers a different task. During session one, participants will be asked to write about their coping strategies to deal with stressors associated with the cancer diagnosis and treatment, as well as future plans for coping with cancer-related stressors; during session two, participants will be asked to write about their deepest feelings and thoughts regarding their experience with breast cancer as well as its impact on their lives; and in session three, participants will be asked to write about positive thoughts and feelings regarding their experience with breast cancer.
  Interventions: Behavioral: Enhanced self-Regulation Condition

INTERVENTIONS:
Behavioral: Self-Regulation Condition
  Arms: Self-regulation condition
Behavioral: Enhanced self-Regulation Condition
  Arms: Enhanced self-regulation condition

SUMMARY:
This study is a randomized controlled trial (RCT) with the aim of determining the cultural sensitivity, feasibility, and effectiveness of an expressive writing intervention for Chinese breast cancer survivors.

DETAILED DESCRIPTION:
The study examines the potential health benefits (i.e., physical health, psychological health, and quality of life) of this expressive writing intervention for Chinese-speaking breast cancer survivors. The study also explores the mechanism through which expressive writing confers health benefits and investigates who will benefit most from the expressive writing intervention. Chinese-speaking breast cancer survivors who have completed primary treatment will be randomly assigned to a control writing condition, a self-regulation condition, or a enhanced self-regulation writing condition. Health outcomes are assessed at baseline, and 1, 3, and 6 months follow-ups. Mixed qualitative-quantitative mixed methods are used to explore the effect of the intervention on health outcomes and explore the mechanisms that explain the benefits of this intervention.

ELIGIBILITY:
Inclusion Criteria:

1) having a breast cancer diagnosis; 2) completing breast cancer surgery within five years; and 3) being comfortable writing and speaking Chinese (i.e. Mandarin or Cantonese)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2012-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in quality of life score as assessed by the Functional Assessment of Cancer Therapy Scale (FACT) | Baseline, 1 month, 3 months, and 6 months follow-ups after the intervention.
  The Functional Assessment of Cancer Therapy Scale (FACT) is a 27-item measure of health-related quality of life (Cella & Tulsky,1993), which assesses perceived life quality in four different facets, including physical well-being (7 items,score range 0 - 28), social well-being (7 items, score range 0 - 28), emotional well-being (6 items, score range 0-24), and functional well-being (7 items, score range 0-28). A higher subscale score indicates better functioning in the corresponding domain.
  Total score is computed by summing up the scores of the four subscales. Total score ranges from 0 to 108. A higher score indicates better quality of life.

SECONDARY OUTCOMES:
Change in posttraumatic stress disorder (PTSD), as assessed by the PTSD Symptom Scale - Self Report version (PSS-SR) | Baseline, 1 month, 3 months, and 6 months follow-ups after the intervention.
  The scale contains 17 items reflecting the Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition -Text Revision (DSM-IV-TR) symptoms of post-traumatic stress disorder (Foa, Riggs, Dancu, & Rothbaum, 1993).
  Score can be reported in terms of total score or the score of the three subscales (Re-experiencing, Avoidance and Hyperarousal).
  The score ranges for the three sub-scales are: Re-experiencing symptoms (5 items, 0-15), Avoidance symptoms (7 items, 0 -21) and Hyperarousal symptoms (5 items, 0-15). Each subscale score is computed by summing up the scores of the corresponding items. For each subscale, a higher score indicates more severe symptoms.
  The total score is computed by summing up the scores of the three subscales. The total score ranges from 0 to 51. A higher score indicated more severe PTSD symptoms.
Change in fatigue as assessed by Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F) | Baseline, 1 month, 3 months, and 6 months follow-ups after the intervention.
  The scale contains 13 items. Total score is computed by summing up the scores of all the 13 items. The total score ranges from 0 to 52. A higher score indicates more severe fatigue symptoms.
Change in depressive symptoms as assessed by Center for Epidemiologic Studies Depression Scale (CES-D). | Baseline, 1 month, 3 months, and 6 months follow-ups after the intervention.
  The scale contains 10 items. Total score is computed by summing up the scores of all the 10 items. Total score ranges from 0 to 30. A higher scores indicates more severe depression symptoms.
Change in anxiety as assessed by Brief Symptom Inventory (BSI)-anxiety dimension | Baseline, 1 month, 3 months, and 6 months follow-ups after the intervention.
  The scale contains 6 items. Total score is computed by summing up the scores of all the 6 items. Total score ranges from 0 - 24. A higher score indicates more severe anxiety symptoms.
Change in physical symptoms as assessed by the Physical Symptoms Checklist | Baseline, 1 month, 3 months, and 6 months follow-ups after the intervention.
  The scale contains 10 items. Total score is computed by summing up the scores of all the 10 items. Total score ranges from 0 - 300. A higher score indicates more severe physical symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Lu, Ph.D., MD, Principal Investigator — University of Houston
Locations (2):
- United States (2):
  - Herald Cancer Association, Los Angeles, California
  - University of Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu Q, Yeung NCY, Tsai W, Kim JHJ. The effects of culturally adapted expressive writing interventions on depressive and anxiety symptoms among Chinese American breast cancer survivors: A randomized controlled trial. Behav Res Ther. 2023 Feb;161:104244. doi: 10.1016/j.brat.2022.104244. Epub 2022 Dec 23. PMID 36592575
- [Derived] Chu Q, Wu IHC, Tang M, Tsoh J, Lu Q. Temporal relationship of posttraumatic stress disorder symptom clusters during and after an expressive writing intervention for Chinese American breast cancer survivors. J Psychosom Res. 2020 Aug;135:110142. doi: 10.1016/j.jpsychores.2020.110142. Epub 2020 May 16. PMID 32485623
- [Derived] Chu Q, Wu IHC, Lu Q. Expressive writing intervention for posttraumatic stress disorder among Chinese American breast cancer survivors: the moderating role of social constraints. Qual Life Res. 2020 Apr;29(4):891-899. doi: 10.1007/s11136-019-02385-5. Epub 2020 Jan 3. PMID 31900761
- [Derived] Lu Q, Gallagher MW, Loh A, Young L. Expressive Writing Intervention Improves Quality of Life Among Chinese-American Breast Cancer Survivors: A Randomized Controlled Trial. Ann Behav Med. 2018 Oct 22;52(11):952-962. doi: 10.1093/abm/kax067. PMID 30346497